CLINICAL TRIAL: NCT03556722
Title: Effectiveness and Tolerability of Repetitive Transcranial Magnetic Stimulation For Preventive Treatment Of Episodic Migraine: A Single Centre, Randomised, Double-Blind, Sham-Controlled Phase 2 Trial
Brief Title: Transcranial Magnetic Stimulation in Episodic Migraine (Magnet-EM)
Acronym: Magnet-EM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Wan Aliaa Wan Sulaiman, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPB/2017/9585500
Record Dates: First submitted 2018-04-27; First posted 2018-06-14 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Migraine
Keywords: Repetitive Transcranial Magnetic Stimulation; Transcranial Doppler; Neuromodulation; Randomized Controlled Trials; Pain; Migraine prophylaxis; Dorsolateral Prefrontal Cortex; Protocol
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment involves two groups of participants. One group receives r-TMS, and the other group receives sham placebo r-TMS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repetitive Transcranial Magnetic Stimulation (Active Comparator): Magstim Rapid-2 (Whitland, Walsh, UK), 70mm Double Air Film Coil given on left dorsolateral prefrontal cortex for five sessions.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation.
- Sham repetitive Transcranial Magnetic Stimulation (Sham Comparator): Magstim Rapid-2 (Whitland, Walsh, UK), 70mm Double Air Film Sham Coil given on left dorsolateral prefrontal cortex for five sessions.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation. — High frequency rTMS on left dorsolateral prefrontal cortex.
  Other Names: rTMS
  Arms: repetitive Transcranial Magnetic Stimulation
Device: Sham rTMS — Sham rTMS without active magnetic coil on left dorsolateral prefrontal cortex.
  Other Names: Placebo
  Arms: Sham repetitive Transcranial Magnetic Stimulation

SUMMARY:
This study will assess the safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) as new preventive treatment of migraine.

DETAILED DESCRIPTION:
Migraine patients according to International Headache Society criteria will be allocated randomly into two treatment arms. One group will receive active rTMS and another group will receive sham rTMS for treatment phase (5 sessions). Assessment will be made at baseline, month 1, month 2 and month 3 post-treatment.

ELIGIBILITY:
Inclusion criteria:

1. Males or females aged 18 to 60 years of age.
2. Subjects fulfilling criteria for episodic migraine as per the Third Edition of The International Headache Society (ICHD-3) for at least 1 year.
3. Frequency of migraine attacks 2-8 times per month with less than 15 headache days per month for at least 3 months prior to screening.
4. Demonstrated compliance with the headache diary during the run-in period by entry of headache data on a minimum of 24/30 days (80% compliance).
5. A signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study including any known and potential risks and available alternative treatments.

Exclusion criteria:

1. Patients with previous history of rTMS treatment.
2. Onset of headache at more than 50-year-old.
3. Headache with red flags symptoms that may suggest organic secondary headaches.
4. Pregnant or lactating women.
5. Patients with contraindications to TMS such as metallic implant and pacemaker based on the Screening 13-item Questionnaire for rTMS candidate.
6. Patients with medical conditions such severe hypertension, infections, malignancy, cardiovascular and cerebrovascular disease, epilepsy degenerative central nervous system diseases, renal failure, hepatic failure, bleeding diathesis and serious mental illness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean monthly migraine days. | Baseline and month 1, 2 and 3 post treatment
  The mean monthly migraine days will be calculated using the monthly migraine days from each of the month of the double-blind treatment phase.

SECONDARY OUTCOMES:
Change from baseline in mean monthly migraine attacks. | Baseline and month 1, 2 and 3 post treatment
  The mean monthly migraine attacks will be calculated using the monthly migraine attack from each of the month of the double-blind treatment phase.
Proportion of subjects with at least a 50% reduction from baseline in mean monthly migraine days. | Baseline and month 1, 2 and 3 post treatment
  Change from baseline in mean monthly pain intensity of migraine attacks. The mean monthly pain intensity will be based on the record of the maximal pain intensity by means of a verbal scale (i.e. 0 =no headache; 1 = mild headache; 2 = moderate headache; 3 = severe headache) prior to taking symptomatic medication.
Frequency and severity of adverse events in response to rTMS. | During treatment and up until 1 month post treatment
  Recorded any adverse events as per Good Clinical Practice Guideline and Declaration of Helsinki.
The Depression Anxiety Stress Scale (DASS 21) score changes in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  Mean score changes from baseline for depression, anxiety and stress category.
The Migraine Disability Assessment Test (MIDAS) score changes in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  Mean score changes from baseline.
The Migraine Specific Questionnaire (MSQ) version 2.1 score changes in migraine patients in response to r-TMS. | Baseline and at month 3 post treatment
  Mean score changes from baseline.
The EQ-5D score changes in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  Mean score changes from baseline.
The Pittsburgh Sleep Quality Index score changes in migraine in response to rTMS. | Baseline and at month 3 post treatment
  Mean score changes from baseline for sleep quality.
The Food Frequency Questionnaire score in migraine patients | Baseline
  Measuring food frequency intake at baseline
The Global Physical Activity Questionnaire score change in migraine in response to rTMS. | Baseline and at month 3 post treatment
  Mean score changes from baseline.
Transcranial Doppler (TCD) pattern changes in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  Mean flow velocity (cm/s).
Electroencephalography (EEG) pattern change in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  EEG pattern differences based on report.
Serum serotonin level in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  Serum serotonin (ng/ml).
Serum beta-endorphin level changes in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  Serum beta endorphin (ng/ml).
Serum Calcitonin gene related peptide (CGRP) level in migraine patients in response to rTMS. | Baseline and at month 3 post treatment
  Serum CGRP (pg/ml).
Satisfaction measures of efficacy, tolerability, safety and expectations of rTMS among the participants. | At month 3 post treatment
  A 5-point, Likert scale will be used to evaluate satisfaction with rTMS in migraine prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Hamidon B. Basri, Study Chair — University Putra Malaysia; Wan Aliaa B. Wan Sulaiman, MRCP, Study Director — Universiti Putra Malaysia; Wan Aliaa B. Wan Sulaiman, MRCP, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- University Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamad Safiai NI, Amir NA, Basri H, Inche Mat LN, Hoo FK, Yusof Khan AHK, Loh WC, Chia PK, Ramachandran V, Mat Din H, Samsudin IN, Fernandez A, Mohamed MH, Ching SM, Hashim HZ, Wan Sulaiman WA. Effectiveness and tolerability of repetitive transcranial magnetic stimulation for preventive treatment of episodic migraine: a single-centre, randomised, double-blind, sham-controlled phase 2 trial (Magnet-EM). Trials. 2020 Nov 11;21(1):923. doi: 10.1186/s13063-020-04832-y. PMID 33176870

DOCUMENTS (3):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03556722/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03556722/SAP_001.pdf
  • Informed Consent Form (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT03556722/ICF_002.pdf